CLINICAL TRIAL: NCT00093028
Title: UARK 2003-35, A Phase III Study of Bortezomib Versus Bortezomib in Two Doses in Combination With Revlimid™ for Patients Relapsing or Progressing on Total Therapy II (UARK 98-026)
Brief Title: Study of Bortezomib and Revlimid™ for Patients Relapsing or Progressing on Total Therapy II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Bart Barlogie, MD, PhD, UAMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UARK 2003-35
Record Dates: First submitted 2004-09-29; First posted 2004-10-01 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Revlimid; bortezomib; CC-5013; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CC-5013 (Revlimid™) — N/A Study Complete
Drug: bortezomib — N/A Study Complete

SUMMARY:
The purpose of this study is

* to find out the effects of treating patients with two new chemotherapy drugs (bortezomib and Revlimid™),
* to study how many patients' myeloma responds to treatment on this study, and how many patients survive after this treatment,
* to learn if a patient's genetic makeup before and after treatment can predict which patients will respond to bortezomib and Revlimid™, and to learn more about how the body responds (gene array studies).

DETAILED DESCRIPTION:
Two new drugs BORTEZOMIB (Velcade®, PS-341) and REVLIMID (CC-5013) have been shown in recent studies to be effective in patients with advanced multiple myeloma. This study is being done to learn more about the best way to administer these drugs, either alone or in combination. Since it is not known at this time which treatment is the best, participants will be placed by chance in one of the three treatment groups:

* BORTEZOMIB alone
* BORTEZOMIB + REVLIMID
* BORTEZOMIB in a lower dose + REVLIMID.

This chance selection process is called randomization and is often used in research studies.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented Multiple Myeloma (MM) previously enrolled on UARK 98-026 with relapsed or progressive disease after at least one autologous transplant.
* Patient has measurable disease in which to capture response, defined as: a. Serum M-protein level > or =1.0 gm/dl (10.0 g/L) measured by serum protein electrophoresis or immunoglobulin electrophoresis b. Urinary M-protein excretion > or =200 mg/24 hrs c. Bone marrow plasmacytosis of > or =30% by bone marrow aspirate and/or biopsy d. Serum Free Light Chains (By the Freelite test) > 2X normal.
* Performance status of < or = 2 as per Zubrod scale, unless PS of 3 based solely on bone pain.
* Patients must have a platelet count > or = 50,000/mm3, and an ANC of at least 1,000/μl.
* Patients must have adequate renal function defined as serum creatinine < or =3.0 mg/dl.
* Patients must have adequate hepatic function defined as serum transaminases and direct bilirubin < or =2 x the upper limit of normal.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Male or female adults of at least 18 years of age.
* Patients must have signed an IRB-approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations

Exclusion Criteria:

* Chemotherapy or radiotherapy received within the previous 2 weeks.
* Not previously enrolled on UARK 98-026.
* Has received either CC-5013 or bortezomib therapy after discontinuing from UARK 98-026.
* Significant neurotoxicity, defined as grade > or = 2 neurotoxicity per NCI Common Toxicity Criteria.
* Platelet count < 50,000/mm3, or ANC < 1,000/μl
* POEMS Syndrome
* Clinically significant hepatic dysfunction as noted by bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association (NYHA) Class III or Class IV heart failure
* Myocardial infarction within the last 6 months.
* Non-secretory MM, unless the patient has measurable lesions on CT, MRI and/or PET.
* Uncontrolled, active infection requiring IV antibiotics.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly controlled hypertension, diabetes mellitus, or other serious or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Pregnant or potential for pregnancy. Women of childbearing potential will have a pregnancy test at screening, and will be required to use a medically approved contraceptive method. Pregnancy testing will be performed prior to administration of each cycle of study drug.
* Breast-feeding women may not participate.
* Known hypersensitivity to thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To find out the effects (good and bad) of treating patients with two new chemotherapy drugs (BORTEZOMIB and REVLIMID). | 24 months

SECONDARY OUTCOMES:
To learn if a patient's genetic makeup before and after treatment can predict which patients will respond to BORTEZOMIB and REVLIMID, and to learn more about how the body responds (gene array studies). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, M.D., Ph.D., Principal Investigator — UAMS Myeloma Institute for Research & Therapy
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu/